CLINICAL TRIAL: NCT04319523
Title: Abnormal Pain Processing in COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, University of Granada, Universidad de Granada
Other Study IDs: DF0087UG
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Pain
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients
- Healthy subjects

SUMMARY:
Dyspnea, cough, and fatigue are the symptoms characteristic of moderate-severe COPD. Within the progression of disease was also reported a prevalence of 34-77% of pain symptoms in these patients. A review observed a higher score in pain intensity/interference associated with multiples pain locations of COPD patients. Pain in chronic diseases may appear to result from abnormalities in pain processing because of the damage and/or inflammation of peripheral structures.

DETAILED DESCRIPTION:
Dyspnea, cough, and fatigue are the symptoms characteristic of moderate-severe COPD. Within the progression of disease was also reported a prevalence of 34-77% of pain symptoms in these patients. A review observed a higher score in pain intensity/interference associated with multiples pain locations of COPD patients. Several studies reported that comorbidities, GOLD grade, and breathlessness may contribute to a higher pain prevalence in COPD patients because of the systemic inflammatory process and lung hyperinflation. Pain in chronic diseases may appear to result from abnormalities in pain processing and alteration of sensitization due to the damage and/or inflammation of peripheral structures.

ELIGIBILITY:
Inclusion Criteria:

* Between 50 and older age
* Accepted to sign the informed consent

Exclusion Criteria:

* comorbidities with a course of chronic pain that interfered with evaluation
* the presence of cognitive impairment to understand the questionnaire

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable COPD patients with a grade III and IV of Global Initiative for Chronic Obstructive Lung Disease (GOLD). Patients were recruited in the pneumology services of San Cecilio and Virgen de las Nieves University Hospitals (Granada, Spain).
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2021-12-03 (Estimated)

PRIMARY OUTCOMES:
Pressure pain thresholds | Baseline
  Pressure pain thresholds (PPT) was used to measure pressure pain sensitivity in muscles with an algometer. With the patient in a seated position, pressure was applied three times at five bilateral points of the body: the distal thumb phalangeal, the gracilis muscle tendon at the inside of the knee, the distal of the middle part of the clavicle, the supraspinous muscle and the trapezius muscle's second portion. When the participant reported that pressure changed to pain, the pressure was stopped, and the mean value was registered.
Temporal summation | Baseline
  Temporal summation (TS) was used to evaluated peripheral sensitization. First, the pressure was applied with gradually increasing pressure until the subject reported pain in the flexor digitorum muscle of each arm. Second, 15 stimuli were applicated to one arm at an interstimulus interval (ISI) of 3 s and then to the other arm at an ISI of 5 s. After a 5 min, the series of stimuli were repeated in reverse order. The evaluation of TS was measured with a standardized numerical scale for rating the magnitude of late sensations experienced during the first, fifth, tenth, and fifteenth stimuli, and 15 and 60 s after the last stimulus in each series to evaluated the temporal summation. The scale ranged from 0 (no pain) to 100 (intolerable pain).

SECONDARY OUTCOMES:
Pain Sensitivity Questionnaire | Baseline
  The Pain Sensitivity Questionnaire (PSQ) measured general pain sensitivity. It consists of 17 items, each describing a daily life situation and asking the patients to rate how painful this situation would be for them on a numeric rating scale ranging from 0 (not painful) to 10 (worst pain imaginable). A major score in the questionnaire a higher pain sensitivity.
Borg scale | Baseline
  The Borg scale was used to assess the dyspnea, which is a comprehensive instrument designed to measure breathlessness in patients with respiratory pathology. Patients rated their dyspnoea from 0 to 10, where 0 represents "no dyspnoea" and 10 represents "maximum dyspnoea." A difference of 0.9 units was considered as the minimal clinically important difference (MCID), according to previous studies in patients with respiratory disease
International Physical Activity Questionnaire | Baseline
  The International Physical Activity Questionnaire (IPAQ) measures total physical activity (MET·minutes·days per week).
Hospital Anxiety and Depression Scale | Baseline
  The HADS is a self-rated questionnaire originally developed for minor depressive symptoms in general medical outpatients. It consists of 14 items, depression (seven items) and anxiety (seven times), each with four choices numbered alphabetically. Each of the subscales' scores ranges from 0 to 21, corresponding to total scores of 0 to 42, with higher scores indicating greater distress.
London Chest Activity of Daily Living | Baseline
  The London Chest Activity of Daily Living (LCADL) was used to assess the impact and severity of breathlessness on ADLs. The LCADL has been used as an outcome measure in COPD. Higher scores reflect greater breathlessness during daily activity and the tool includes an anchor question identifying an individual's overall perception of the impact of breathlessness on their daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Andalusia, Spain